CLINICAL TRIAL: NCT04246047
Title: DREAMM 7: A Multicenter, Open-Label, Randomized Phase III Study to Evaluate the Efficacy and Safety of the Combination of Belantamab Mafodotin, Bortezomib, and Dexamethasone (B-Vd) Compared With the Combination of Daratumumab, Bortezomib and Dexamethasone (D-Vd) in Participants With Relapsed/Refractory Multiple Myeloma
Brief Title: Evaluation of Efficacy and Safety of Belantamab Mafodotin, Bortezomib and Dexamethasone Versus Daratumumab, Bortezomib and Dexamethasone in Participants With Relapsed/Refractory Multiple Myeloma
Acronym: DREAMM 7
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207503; 2018-003993-29 (EudraCT Number)
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Multiple Myeloma
Keywords: Global Cohort; Belantamab mafodotin; Relapsed/refractory multiple myeloma; Daratumumab; Bortezomib; Dexamethasone; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belantamab mafodotin and Bortezomib plus Dexamethasone (Arm A) (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Dexamethasone
- Daratumumab and Bortezomib plus Dexamethasone (Arm B) (Active Comparator)
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab mafodotin — Humanized anti-B-cell maturation antigen (BCMA) antibody/drug conjugate
  Arms: Belantamab mafodotin and Bortezomib plus Dexamethasone (Arm A)
Drug: Daratumumab — Anti-cluster of differentiation 38 [CD-38] monoclonal antibody
  Arms: Daratumumab and Bortezomib plus Dexamethasone (Arm B)
Drug: Bortezomib — Proteasome Inhibitor
Drug: Dexamethasone — Synthetic glucocorticoid with anti-tumor activity

SUMMARY:
This is a Phase 3, randomized, open-label study designed to evaluate safety and efficacy of belantamab mafodotin in combination with bortezomib/dexamethasone (Arm A) versus daratumumab in combination with bortezomib/dexamethasone (Arm B) in the participants with relapsed recurrent multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma as defined by the International Myeloma Working Group (IMWG) criteria.
* Previously treated with at least 1 prior line of multiple myeloma (MM) therapy, and must have documented disease progression during or after their most recent therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Must have at least 1 aspect of measurable disease, defined as one of the following;

  1. Urine M-protein excretion >=200 mg per 24-hour, or
  2. Serum M-protein concentration >=0.5 grams per deciliter (g/dL), or
  3. Serum free light chain (FLC) assay: involved FLC level >=10 mg per dL (>=100 mg per liter) and an abnormal serum free light chain ratio (<0.26 or >1.65).
* All prior treatment-related toxicities (defined by National Cancer Institute Common Toxicity Criteria for Adverse Events [NCI-CTCAE] version 5.0) must be <=Grade 1 at the time of enrollment, except for alopecia.
* Adequate organ function

Exclusion Criteria:

* Intolerant to daratumumab.
* Refractory to daratumumab or any other anti-CD38 therapy (defined as progressive disease during treatment with anti-CD38 therapy, or within 60 days of completing that treatment).
* Intolerant to bortezomib, or refractory to bortezomib (defined as progressive disease during treatment with a bortezomib-containing regimen of 1.3 mg/m^2 twice weekly, or within 60 days of completing that treatment). Note: participants with progressive disease during treatment with a weekly bortezomib regimen are allowed.
* Ongoing Grade 2 or higher peripheral neuropathy or neuropathic pain.
* Prior treatment with anti-B-cell maturation antigen (anti-BCMA) therapy.
* Prior allogenic stem cell transplant.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions, including renal, liver, cardiovascular, or certain prior malignancies.
* Corneal epithelial disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2026-06-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (129):
- United States (6):
  - GSK Investigational Site, Yuma, Arizona
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fairfield, Connecticut
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Roanoke, Virginia
- Australia (13):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Waratah, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Benowa, Queensland
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Ashford, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
  - GSK Investigational Site, Nedlands, Western Australia
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Roeselare
- Brazil (6):
  - GSK Investigational Site, Florianópolis
  - GSK Investigational Site, Joinville
  - GSK Investigational Site, Natal
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- China (10):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shenyang
  - GSK Investigational Site, Suzhou
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Zhengzhou
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
- France (5):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rennes
- Germany (6):
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Düsseldorf
  - GSK Investigational Site, Jena
  - GSK Investigational Site, München
  - GSK Investigational Site, Ulm
  - GSK Investigational Site, Würzburg
- Greece (3):
  - GSK Investigational Site, Alexandroupoli
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
- Israel (4):
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Tel Aviv
  - GSK Investigational Site, Tel Litwinsky
- Italy (10):
  - GSK Investigational Site, Bergamo
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Catania
  - GSK Investigational Site, Meldola FC
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Ravenna
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Siena
  - GSK Investigational Site, Torino
- Japan (13):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Aomori
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
- Netherlands (2):
  - GSK Investigational Site, Dordrecht
  - GSK Investigational Site, Groningen
- New Zealand (4):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Takapuna Auckland
  - GSK Investigational Site, Wellington
- Poland (7):
  - GSK Investigational Site, Chorzów
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Nowy Sącz
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- Russia (7):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Ufa
- South Korea (4):
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Ulsan
- Spain (10):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Gijón
  - GSK Investigational Site, L'Hospitalet de Llobrega
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, MOstoles Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, PamplonaNavarra
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Salamanca
- United Kingdom (7):
  - GSK Investigational Site, Bournemouth
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, London
  - GSK Investigational Site, Stoke-on-Trent
  - GSK Investigational Site, Sutton

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

REFERENCES:
- [Derived] Mateos MV, Trudel S, Quach H, Robak P, Beksac M, Pour L, Hus M, Kim K, Zherebtsova V, Delimpasi S, Jelinek T, Ward C, Ho PJ, Vorobyev V, Pitombeira de Lacerda M, Aparecida-Martinez G, Spicka I, Radocha J, Cavo M, Cerchione C, Fu C, Suzuki K, Rogers R, Phillips-Jones A, Wang Z, Baig H, Wilkes J, Zhou XL, Lewis E, Eccersley L, Sule N, Paka P, Opalinska JB, Mukhopadhyay P, Hungria V, Dimopoulos MA. Modification of belantamab mafodotin dosing to balance efficacy and tolerability in the DREAMM-7 and DREAMM-8 trials. Blood Adv. 2025 Nov 25;9(22):5708-5719. doi: 10.1182/bloodadvances.2025016949. PMID 40763276
- [Derived] Hungria V, Robak P, Hus M, Zherebtsova V, Ward C, Ho PJ, Hajek R, Kim K, Grosicki S, Sia H, Bryant A, Pitombeira de Lacerda M, Martinez GA, Sureda Balari A, Sandhu I, Cerchione C, Ganly P, Dimopoulos MA, Fu C, Garg M, Abdallah AO, Gatt ME, Oriol Rocafiguera A, Cavo M, Rifkin R, Fujisaki T, Mielnik M, Ficek J, Mantero A, Pirooz N, Varghese S, Lee J, McKeown A, Rogers R, Baig H, Eccersley L, Roy-Ghanta S, Mukhopadhyay P, Nielsen J, Opalinska J, Mateos MV; DREAMM-7 study investigators. Belantamab mafodotin plus bortezomib and dexamethasone in patients with relapsed or refractory multiple myeloma (DREAMM-7): updated overall survival analysis from a global, randomised, open-label, phase 3 trial. Lancet Oncol. 2025 Aug;26(8):1067-1080. doi: 10.1016/S1470-2045(25)00330-4. Epub 2025 Jul 15. PMID 40680754
- [Derived] Hungria V, Hus M, Fu C, Zherebtsova V, Ward C, Ho PJ, Mikulski D, Muronova L, Cerchione C, Loubert A, Bunod L, M'Hari M, Pirooz N, Rogers R, Lin CP, Roy-Ghanta S, Opalinska JB, Purser M, McKeown A, McNamara S, Baig H, Eccersley L, Pompilus F, Mateos MV; DREAMM-7 trial study group. Patient-reported outcomes with belantamab mafodotin, bortezomib, and dexamethasone versus daratumumab, bortezomib, and dexamethasone in patients with relapsed or refractory multiple myeloma (DREAMM-7): results from a phase 3, open-label, randomised controlled trial. Lancet Haematol. 2025 Aug;12(8):e599-e610. doi: 10.1016/S2352-3026(25)00163-2. Epub 2025 Jul 15. PMID 40680752
- [Derived] Hungria V, Robak P, Hus M, Zherebtsova V, Ward C, Ho PJ, Ribas de Almeida AC, Hajek R, Kim K, Grosicki S, Sia H, Bryant A, Pitombeira de Lacerda M, Aparecida Martinez G, Sureda Balari AM, Sandhu I, Cerchione C, Ganly P, Dimopoulos M, Fu C, Garg M, Abdallah AO, Oriol A, Gatt ME, Cavo M, Rifkin R, Fujisaki T, Mielnik M, Pirooz N, McKeown A, McNamara S, Zhou X, Nichols M, Lewis E, Rogers R, Baig H, Eccersley L, Roy-Ghanta S, Opalinska J, Mateos MV; DREAMM-7 Investigators. Belantamab Mafodotin, Bortezomib, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2024 Aug 1;391(5):393-407. doi: 10.1056/NEJMoa2405090. Epub 2024 Jun 1. PMID 38828933

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results presented are until the primary completion date. Additional results will be provided within a year of study completion.
Groups:
- Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex): Participants with Relapsed/Refractory Multiple Myeloma (RRMM) received intravenous (IV) infusion of 2.5 milligram (mg)/kilogram (kg) belantamab mafodotin on Day 1 of each 21-day Cycle until disease progression, intolerable toxicity, death, informed consent withdrawal, or study end, whichever comes first in combination with 1.3 mg/meter^2 (m^2) Bor administered subcutaneously (SC) once daily on Days 1, 4, 8 and 11 of each 21-day cycle along with 20 mg Dex via oral tablet or IV infusion once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle for a total of 8 cycles.
- Daratumumab + Bor + Dex: Participants with RRMM received 16 mg/kg Daratumumab IV infusion once weekly of each 21-day cycle in Cycle 1 to Cycle 3; once every 3 weeks on Day 1 of each 21-day cycle in Cycle 4 to Cycle 8; and once every 4 weeks on day 1 of each 28-day cycle from cycle 9 onwards until disease progression, intolerable toxicity, death, informed consent withdrawal, or study end, whichever comes first in combination with 1.3 mg/m^2 Bor administered SC once daily on Days 1, 4, 8 and 11 of each 21-day cycle along with 20 mg Dex oral tablet or IV infusion once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle for a total of 8 cycles.
Period: Overall Study
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex
Started (Intent-to-Treat (ITT) Population included of all randomized participants whether or not randomized treatment was administered.) | 243 | 251
Safety Population (Participants randomized who took at least 1 dose of study treatment.) | 242 | 246
Completed | 0 | 0
Not Completed | 243 | 251
Not completed — Death | 50 | 77
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 4 | 10
Not completed — Withdrawal by Subject | 19 | 26
Not completed — Ongoing | 169 | 135

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex | Total
Number analyzed (Participants) | 243 | 251 | 494
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 64.5 (9.47) | 63.6 (10.11) | 64.0 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 107 | 222
  Male | 128 | 144 | 272
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 41 | 71
  Not Hispanic or Latino | 213 | 208 | 421
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as time from randomization until earliest date of disease progression (PD), determined by Independent Review Committee (IRC), according to the International Myeloma Working Group (IMWG) Response Criteria, or death due to any cause. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5 grams per deciliter {g/dL}]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200 milligrams per 24 hours {mg/24h}]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved serum free light chains (sFLC) levels [absolute increase >10mg/dL]; appearance of new lesion,>=50% increase from nadir in Sum of the products of the maximal perpendicular diameters of measured lesions (SPD) of >1 lesion, or >=50% increase in longest diameter of previous lesion >1 centimeter (cm) in short axis.
Time Frame: Up to approximately 41 months
Population: Intent-to-Treat (ITT) Population included of all randomized participants whether or not randomized treatment was administered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex
Number analyzed (Participants) | 243 | 251
Months | 36.6 [28.4 to NA] — NA indicates the upper limit of 95% CI was not able to be estimated due to length of follow-up in assessing the number of events. | 13.4 [11.1 to 17.5]
Statistical Analysis 1: Comparison: Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) vs Daratumumab + Bor + Dex; Test type: Superiority; p < 0.00001, one-sided stratified log-rank; Hazard Ratio (HR) = 0.41, 95% CI [0.31 to 0.53] — Hazard ratio was estimated using a Cox Proportional Hazards model stratified by the number of lines of prior therapy, prior bortezomib and revised international staging system (R-ISS) at screening, with a covariate of treatment

2. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as percentage of participants with a confirmed complete response or better.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as percentage of participants with a confirmed partial response or better.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as percentage of participants with a confirmed minimal response (MR) or better
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

5. Secondary Outcome: Duration of Response (DoR)
Description: DOR is defined as time from first documented evidence of partial response or better until first documented progression or death, whichever occurs first.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

6. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as time from the date of randomization and the first documented evidence of response (PR or better) among participants who achieve partial response or better.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

7. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as time from the date of randomization until the earliest date of documented date of disease progression or death, whichever occurs first.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from the date of randomization until the date of death due to any cause.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

9. Secondary Outcome: Progression-free Survival on Subsequent Line of Therapy (PFS2)
Description: Progression-free survival on subsequent line of therapy is defined as time from randomization to disease progression after initiation of new anti-myeloma therapy or death from any cause, whichever occurs first. If disease progression after new antimyeloma therapy cannot be measured, a PFS event is defined as the date of discontinuation of new anti-myeloma therapy, or death from any cause, whichever is earlier.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

10. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate
Description: Minimal Residual Disease (MRD) negativity rate is defined as the percentage of participants who are MRD negative status by next generation sequencing (NGS).
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples will be collected for the analysis of hematology parameters.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Chemistry
Description: Blood samples will be collected for the analysis of clinical chemistry parameters.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Urine Dipstick
Description: Urine samples will be collected for the urine dipstick analysis.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

15. Secondary Outcome: Number of Participants With Abnormal Ocular Findings on Ophthalmic Examination
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

16. Secondary Outcome: Plasma Concentrations of Belantamab Mafodotin (Total Antibody) at Indicated Time Points
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

17. Secondary Outcome: Plasma Concentrations of Belantamab Mafodotin (ADC) at Indicated Time Points
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

18. Secondary Outcome: Plasma Concentrations of Monomethyl Auristatin-F With a Cysteine Linker (Cys-mcMMAF) at Indicated Time Points
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

19. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples collected for the analysis of the presence of ADAs using validated immunoassays. All samples will be tested in screening assay, and positive samples will be further characterized for antibody titers.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

20. Secondary Outcome: Titers of ADAs Against Belantamab Mafodotin
Description: Serum samples collected for the analysis of the presence of ADAs using validated immunoassays. All samples will be to be further tested in screening assay, and positive samples will be further to be characterized for antibody titers.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

21. Secondary Outcome: Number of Participants With Maximum Post-baseline Change From Baseline in Individual Items of Patient-Reported Outcome Version of the Common Term Criteria for Adverse Events (PRO-CTCAE)
Description: The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicity in participants on cancer clinical trials. The PRO-CTCAE includes an item library of 124 items representing 78 symptomatic toxicities drawn from the CTCAE.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

22. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQoL) as Measured by EuropeanOrganization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core Module (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 includes 30-items with single and multi-item scales. These included five functional scales (physical functioning [PF], role functioning [RF], cognitive functioning [CF], emotional functioning [EF] and social functioning [SF]), three symptom scales (fatigue, pain and nausea/vomiting [N/V]), a global health status (GHS)/ Quality-of-Life (QoL) scale, and six single items (constipation, diarrhoea, insomnia, dyspnoea, appetite loss [AL] and financial difficulties [FD]). Response options are 1 to 4. Scores were averaged and transformed to 0 to 100, a high score for functional scales/ GHS/QoL represent better functioning ability or health-related quality-of-life (HRQoL), whereas a high score for symptom scales/ single items represent significant symptomatology. Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

23. Secondary Outcome: Change From Baseline in HRQoL as Measured by EORTC IL52
Description: The EORTC Quality of Life Questionnaire 20-item Multiple Myeloma module (QLQMY20) is a supplement to the QLQ-C30 instrument used in participants with multiple myeloma. For the EORTC IL52, disease symptoms domain of the QLQ-MY20 will be used for bone aches or pain, back pain, hip pain, arm or shoulder pain, chest pain, and pain increasing with activity. The individual component scores in the disease symptom domain are averaged and transformed linearly to a score ranging from 0 to100. A high score for disease symptoms represents a high level of symptomatology or problems. A high score represents a high/healthy level of functioning.
Time Frame: Up to 73 months
Reporting Status: Not Posted, anticipated posting 2027-06

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to approximately 41 months. The results presented are until the primary completion date. Additional results will be provided within a year of study completion.
Description: Safety population included all randomized participants who took at least 1 dose of study treatment.
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex
All-Cause Mortality (participants affected / at risk) | 50/242 | 77/246
Serious Adverse Events (participants affected / at risk) | 121/242 | 90/246
Other Adverse Events (participants affected / at risk) | 238/242 | 239/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) (N=242) | Daratumumab + Bor + Dex (N=246)
Pneumonia (Infections and infestations) | 27 (27) | 10 (13)
COVID-19 (Infections and infestations) | 11 (11) | 10 (10)
COVID-19 pneumonia (Infections and infestations) | 8 (8) | 8 (8)
Sepsis (Infections and infestations) | 3 (3) | 4 (4)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 1 (1)
Atypical pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0)
Leishmaniasis (Infections and infestations) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 12 (12) | 9 (9)
Chest pain (General disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Injection site extravasation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peroneal nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (11) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 3 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 4 (4) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 4 (5) | 3 (4)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of conjunctiva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 3 (5) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) (N=242) | Daratumumab + Bor + Dex (N=246)
Thrombocytopenia (Blood and lymphatic system disorders) | 167 (501) | 122 (269)
Anaemia (Blood and lymphatic system disorders) | 45 (66) | 64 (110)
Neutropenia (Blood and lymphatic system disorders) | 34 (83) | 27 (51)
Lymphopenia (Blood and lymphatic system disorders) | 21 (44) | 23 (38)
Leukopenia (Blood and lymphatic system disorders) | 14 (42) | 10 (17)
Peripheral sensory neuropathy (Nervous system disorders) | 61 (81) | 51 (68)
Neuropathy peripheral (Nervous system disorders) | 50 (59) | 55 (70)
Dizziness (Nervous system disorders) | 21 (24) | 19 (20)
Headache (Nervous system disorders) | 21 (25) | 18 (20)
Polyneuropathy (Nervous system disorders) | 15 (17) | 13 (14)
Paraesthesia (Nervous system disorders) | 14 (16) | 13 (14)
Diarrhoea (Gastrointestinal disorders) | 76 (109) | 77 (119)
Constipation (Gastrointestinal disorders) | 46 (53) | 56 (72)
Nausea (Gastrointestinal disorders) | 39 (43) | 30 (40)
Vomiting (Gastrointestinal disorders) | 14 (16) | 24 (31)
Abdominal pain (Gastrointestinal disorders) | 19 (23) | 12 (13)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 14 (16)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 13 (13)
Vision blurred (Eye disorders) | 160 (471) | 25 (32)
Dry eye (Eye disorders) | 123 (279) | 17 (18)
Photophobia (Eye disorders) | 114 (247) | 6 (7)
Eye irritation (Eye disorders) | 103 (250) | 13 (17)
Foreign body sensation in eyes (Eye disorders) | 106 (253) | 10 (14)
Eye pain (Eye disorders) | 77 (139) | 8 (10)
Cataract (Eye disorders) | 48 (66) | 25 (30)
Visual impairment (Eye disorders) | 26 (57) | 4 (6)
Lacrimation increased (Eye disorders) | 21 (44) | 7 (7)
Visual acuity reduced (Eye disorders) | 14 (20) | 5 (5)
COVID-19 (Infections and infestations) | 53 (60) | 46 (48)
Upper respiratory tract infection (Infections and infestations) | 48 (80) | 49 (72)
Pneumonia (Infections and infestations) | 29 (35) | 15 (17)
Urinary tract infection (Infections and infestations) | 21 (26) | 20 (28)
Bronchitis (Infections and infestations) | 22 (29) | 13 (15)
Platelet count decreased (Investigations) | 51 (98) | 40 (87)
Alanine aminotransferase increased (Investigations) | 47 (69) | 29 (40)
Aspartate aminotransferase increased (Investigations) | 37 (59) | 13 (20)
Gamma-glutamyltransferase increased (Investigations) | 36 (44) | 11 (14)
Blood lactate dehydrogenase increased (Investigations) | 28 (55) | 8 (16)
Weight decreased (Investigations) | 15 (15) | 9 (10)
Lymphocyte count decreased (Investigations) | 9 (16) | 14 (33)
Neutrophil count decreased (Investigations) | 9 (14) | 14 (23)
Blood creatinine increased (Investigations) | 6 (6) | 13 (22)
Blood alkaline phosphatase increased (Investigations) | 13 (15) | 4 (5)
Fatigue (General disorders) | 47 (52) | 48 (57)
Pyrexia (General disorders) | 35 (44) | 19 (24)
Oedema peripheral (General disorders) | 26 (29) | 22 (24)
Asthenia (General disorders) | 19 (27) | 22 (25)
Hypokalaemia (Metabolism and nutrition disorders) | 27 (38) | 26 (47)
Decreased appetite (Metabolism and nutrition disorders) | 23 (26) | 22 (22)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (21) | 29 (39)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (11) | 17 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (23) | 36 (40)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (27) | 25 (34)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (15) | 25 (30)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (34) | 33 (40)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 23 (26)
Insomnia (Psychiatric disorders) | 38 (42) | 47 (55)
Hypertension (Vascular disorders) | 28 (30) | 19 (19)
Infusion related reaction (Injury, poisoning and procedural complications) | 8 (8) | 38 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT04246047/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT04246047/SAP_001.pdf